CLINICAL TRIAL: NCT04108559
Title: Comparison of The Surgical Drain Placement With Use of Kinesiologic Tape on Postoperative Pain, Swelling and Trismus in Impacted Mandibular Third Molar Surgery
Brief Title: Comparison of The Surgical Drain Placement With Use of Kinesiologic Tape
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Dilek Menziletoglu, Principle Investigator, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NEU4
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-08

CONDITIONS: Impacted Third Molar Tooth
Keywords: Kinesiology tape; Surgical drain; Pain; Swelling; Trismus
MeSH Terms: conditions — Pain; Trismus | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesiologic Tape Group (Experimental): After the routine impacted third molar surgery, the kinesiologic tape will be prepared individually for each patient; it will be cut into three equal strips (approximately 1.6 cm in width) and placed between the clavicle and the tragus-commissura line. Kinesiologic tape will be removed on the second postoperative day, and all sutures on will be removed on 7. postoperative day.
  Interventions: Procedure: Kinesiologic Tape Group
- Surgical Drain Group (Experimental): After routine impacted third molar surgery, plastic non-customised drain tube (2-cm long, 2-mm diameter) will be inserted into a vertical incision between the first and second molars and sutured to the vestibular mucosa.
  Interventions: Procedure: Drain Group
- Control Group (Placebo Comparator): Routine third molar extraction will be performed. No extra procedures will be done after surgery.
  Interventions: Other: Control Group

INTERVENTIONS:
Procedure: Kinesiologic Tape Group — A mucoperiosteal flap will be raised, a conventional rotary handpiece will be used under irrigation for removing the third molar.Primary wound closure will be accomplished using 3-0 silk sutures.The kinesiologic tape will be prepared individually for each patient; it will be cut into three equal strips (approximately 1.6 cm in width) and placed between the clavicle and the tragus-commissura line. The patients will be invited after one week for removing the sutures.
  Arms: Kinesiologic Tape Group
Procedure: Drain Group — A mucoperiosteal flap will be raised, a conventional rotary handpiece will be used under irrigation for removing the third molar.Primary wound closure will be accomplished using 3-0 silk sutures. A plastic non-customised drain tube (2-cm long, 2-mm diameter) will be inserted into a vertical incision between the first and second molars and sutured to the vestibular mucosa. The patients will be invited after one week for removing the sutures.
  Arms: Surgical Drain Group
Other: Control Group — Routine third molar extraction will be performed. No extra procedures will be done after surgery.
  Arms: Control Group

SUMMARY:
The investigator's purpose was to compare the effects of the surgical drain and kinesiologic tape applications on postoperative morbidity after mandibular third molar surgery.

DETAILED DESCRIPTION:
A total of 90 patients will be scheduled for impacted third molar surgery. The patients will be divided into 3 groups.All surgeries will be carried out by the same surgeon. Group A will be treated with kinesiologic tape, Group B will be treated with a surgical drainage tube and Group C will be control group. After surgery in control group, routine surgical extraction will be performed.The investigators will compare postoperative pain, swelling, trismus and patients' comfort.

The duration of each procedure from the start of the incision to the time of last suture placement will be noted.

Patients are recalled on days 2, 7, 14 postoperative pain, facial swelling, maximum mouth opening, wound dehiscence. For the assesment of the pain, visual analog scale will be used. For the swelling evaluation, measurement will be done from the different three region on the face:

* Tragus-Pogonion
* Tragus-Labial Commissura
* Angulus Mandible-Lateral canthus

Maximum mouth opening will be noted before and after (one week later) the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 of age,
* Asymptomatic bilateral mesioangular impacted mandibular third molar (Pell and Gregory class II, position B)
* Fully covered with mucosa and bone

Exclusion Criteria:

* Alcohol abuse,
* Smoking,
* Pregnancy,
* No allergy
* Presence of acute severe periodontitis.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Swelling will be assessed using paper ruler. Tragus-Pogonion Tragus-Labial Commissura Angulus Mandible-Lateral canthus. | Up to 1week
  Swelling measurement will be done from the different three region on the face. Tragus-Pogonion Tragus-Labial Commissura Angulus Mandible-Lateral canthus. The swelling measurement will be done preoperatively, postoperative 2nd day, 7th day after the surgery.
Pain will be assessed using a visual analogue scale. | Up to 1week
  The level of postoperative pain will be evaluated using a 10-cm visual analogue scale , with zero representing no pain and 10 representing excruciating pain. Pain measurement will be done everyday in one week after the surgery.
Trismus will be evaluated using a caliper at maximum mouth opening. | Up to 1week
  Trismus will be assessed by measuring the maximum interincisal opening (in millimetres) - the distance between the incisal margin of the upper and lower central incisors. Trismus measurement will be done preoperatively, postoperative 2nd day, 7th day after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menziletoglu, Dr, Principal Investigator — Necmettin Erbakan University; Bozkurt Ku Isik, Prof Dr, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No